CLINICAL TRIAL: NCT00229866
Title: Feeding After Neonatal Surgery Chart Review
Brief Title: Feeding After Neonate Surgery Review
Status: Terminated | Type: Observational
Why Stopped: sufficient data gathered for study conclusion
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-072
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Congenital Disorders
Keywords: newborn; pediatric health; Feeding difficulty; discharge with a NG tube; G-tube placement; Nissen fundoplication
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to determine what factors, if any, lead to delayed feeding, discharge with a NG tube, G-tube placement or Nissen fundoplication.

DETAILED DESCRIPTION:
The purpose is to determine what factors, if any, lead to delayed feeding, discharge with a NG tube, G-tube placement or Nissen fundoplication. Will review the newborn database (Lumedx as most interested in those children who have never been fed prior to their cardiac surgery. The medical charts will be reviewed at Children's Healthcare of Atlanta at Egleston Hospital. Approximately 90 charts will be reviewed for newborns undergoing surgery in the 2003 calendar year.

The factors that will be reviewed are pre-op feeding regimen, diagnosis, single vs two ventricle, open vs closed heart procedure, length of bypass, level of hypothermia, circulatory arrest, presence of TEE probe and post-op ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who undergo cardiac surgery

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates who undergo cardiac surgery
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2005-08; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States